CLINICAL TRIAL: NCT05756101
Title: General Scientific Research Project of Zhejiang Provincial Department of Education
Brief Title: Application of New Restraint Instruments in Safety Management of Patients After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: 2022-0916
Record Dates: First submitted 2023-02-07; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-01

CONDITIONS: After Cardiac Surgery
Keywords: Restraints；Postoperative patients；Security management
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Sponge restraint belt, restraint method: adjust the fixed wrist strap according to the diameter of the patient's hand (foot) wrist, and then circle the fixed strap around the wrist strap, one end is pierced through the strap hole without knots, and the two ends of the fixed strap are fixed on both sides of the bed as needed.
  Interventions: Device: Research on the application of novel restraint devices in postoperative patient safety management in cardiac surgery
- Experimental group (Experimental): A new type of restraint device, which is an adjustable protective restraint device (patent number ZL202020155913.1), including upper fixation bracket I, upper fixation bracket II, lower fixation bracket I, lower fixation bracket II and gloves; The plurality of fixed brackets are provided with breathable holes and breathable cotton is placed to increase air permeability and comfort. Place the patient's elbow joint on top of the lower fixation bracket I and II, and then install and connect the upper fixation bracket I and the upper fixation bracket 2 through the upper and lower tightening belts, and adjust their tightness; The upper and lower fixed bracket connections are adjustment module 1 and adjustment module 2, forming a detachable and rotating connection within a certain angle range to adjust the angle of elbow joint movement of the patient; The patient's hand is made by wearing gloves with a grip ball on the palm surface.
  Interventions: Device: Research on the application of novel restraint devices in postoperative patient safety management in cardiac surgery

INTERVENTIONS:
Device: Research on the application of novel restraint devices in postoperative patient safety management in cardiac surgery — According to the individual characteristics of ICU patients and the needs of patients, a new type of restraint device was innovatively made and the effectiveness and safety of the new restraint device were studied, which provided clinical reference and theoretical basis for standardizing postoperative patient restraint.

SUMMARY:
Restraint devices refer to various devices that restrict the activities of the body or a certain part of the body for patients who self-injure or may harm others, so as to maintain the safety of patients and ensure the smooth progress of treatment and care. The essence of restraint devices is to limit patient movement in order to reduce the risk of unexpected adverse events. With the in-depth implementation of high-quality nursing services, nurses have also paid more and more attention to restraint nursing and developed a variety of restraint tools. Common restraints include bed rails, wrist or ankle restraint straps, restraint vests, shoulder or belt-style restraint straps, mittens, etc. According to the limitations of traditional restraints, Deng Wandi et al. innovatively produced double safety restraint belts, racket gloves and safety vests, and the research results showed that innovative new restraint devices can effectively reduce the psychological pressure of nurses and improve the complications caused by restraint. According to the characteristics of critically ill patients, Xu Yan et al. innovatively produced a three-piece set of safety protection restraint equipment on the basis of the original restraint equipment, which is composed of a safety restraint vest, restraint gloves and knee restraint belt, and the research results show that the new restraint device can effectively reduce the adverse events caused by restraint and improve the satisfaction of family members.

In view of the above problems, our department has developed a new protective restraint device for the protective restraint of postoperative intubated patients, and summarizes the nursing experience to provide clinical reference and theoretical basis for standardizing postoperative patient constraints. The project is now a general scientific research project of Zhejiang Provincial Department of Education, the project name is "Application Research of New Restraint Devices in Postoperative Patient Safety Management in Cardiac Surgery", and the funding source is self-financing.According to the individual characteristics of ICU patients and the needs of patients, a new type of restraint device was innovatively made and the effectiveness and safety of the new restraint device were studied, which provided clinical reference and theoretical basis for standardizing postoperative patient restraint.

DETAILED DESCRIPTION:
The study set up control group and experimental group. The control group used sponge restraint belt full name: Medical Care Pad, specifications for: limb restraint belt (Limb Belt Type) . Manufacturer: Shaoxing City, Zhuji City, Zhejiang province, southern Shuda medical supplies factory. The experimental group used an adjustable protective restraint device, including an upper fixing bracket, an upper fixing bracket, a lower fixing bracket, a lower fixing bracket and gloves Air permeability holes are arranged on the fixed supports and air permeability cotton is arranged to increase air permeability and comfort. The elbow joint of the patient was placed on the upper and the lower fixing bracket, and then connected to the upper fixing bracket and the upper fixing bracket through the upper and lower tightening belts, respectively, and the tightness of the upper and lower fixing bracket was adjusted The joint of the upper and lower fixed bracket is the adjustment module one and the adjustment module two, forming a detachable rotational connection in a certain angle range to adjust the patient's elbow joint movement angle; The patient's hand is equipped with a glove with a gripping ball on the palm surface.The national standard for products conforms to GB/T 16886.10-2017/ISO 10993-10:2010, biological evaluation of medical devices, part 10: standards for stimulation and skin sensitization tests.

ELIGIBILITY:
Inclusion Criteria:

* (1) Elective surgery patients, age ≥ 18 years old; (2) Clear preoperative consciousness and no communication barriers; (3) The surgical method is open-heart surgery under intravenous or inhalation general anesthesia; (4) During ICU treatment, there is endotracheal intubation; (5) Before restraint, there is no joint dysfunction, edema, skin damage, etc. in the site to be restrained, and the peripheral circulation is good; (6) Informed consent and voluntary participation in this study.

Exclusion Criteria:

* (1) history of psychiatric illness; (2) Have bleeding tendency or skin diseases; (3) Voluntarily abandon treatment or die halfway.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Unplanned extubation rate | This study began with the patient's postoperative use of the protective restraint tool and ended with the removal of the endotracheal intubation to release the protective restraint.No more than a month.
  Unplanned extubation includes extubation without the consent of the healthcare provider; b. The pipeline slips due to various reasons; c. Due to catheter quality problems and catheter blockage, it is necessary to extubate in advance. Unplanned extubation rate = number of unplanned extubation cases in the same period / total number of ICU hospitalizations in the statistical period× 100%.

DOCUMENTS (1):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT05756101/Prot_000.pdf